CLINICAL TRIAL: NCT02031900
Title: High Resolution Optical Imaging of the Esophagus Using the NvisionVLE™ Imaging System
Status: Completed | Type: Observational
Sponsor: NinePoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-01
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Undergoing Esophagogastroduodenoscopy (EGD)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Undergoing EGD
  Interventions: Device: NvisionVLE Imaging System: NvisionVLE Imaging Console, NvisionVLE Optical Probe and Inflation Accessory Kit

INTERVENTIONS:
Device: NvisionVLE Imaging System: NvisionVLE Imaging Console, NvisionVLE Optical Probe and Inflation Accessory Kit — The NvisionVLE Imaging System is indicated for use as an imaging tool in the evaluation of human tissue microstructure, including esophageal tissue microstructure, by providing two-dimensional, cross-sectional, real-time depth visualization.

SUMMARY:
This is a single center, single arm, open label observational trial of patients undergoing EGD. The primary objective of this clinical trial is to evaluate the ability of physicians to position the NvisionVLE Optical Probe to acquire an image of an area of the esophagus to identify and discriminate abnormal areas of tissue from normal.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years.
* Patients presenting for an EGD.
* Ability to provide written, informed consent.
* Females who are able to become pregnant, are willing to take a pregnancy test.

Exclusion Criteria:

* Patients on anticoagulation undergoing high risk procedures in accordance to ASGE guideline for the management of antithrombotic agents for endoscopic procedures (2009)*.
* Patients with esophageal varices that preclude biopsies.
* Presence of an esophageal mass that precludes full distention of the balloon from the NvisionVLE catheter.
* Patients with esophageal strictures that would prevent adequate expansion of the balloon from the NvisionVLE catheter.
* Patients with known inflammatory disease, esophageal tears or ulcers, which prohibit full distention of the balloon from the NvisionVLE catheter.
* Patients with known eosinophilic esophagitis.
* Patients that are pregnant.
* Patients with a history of hemostasis disorders**.

  * Patients on anticoagulation undergoing low risk procedures are not excluded. ** Hemostasis disorders will include, but will not be limited to: patients with hemophilia or other congenitally acquired clotting factor deficiencies, patients with cirrhosis with coagulopathy, patients known to have thrombocytopenia (<100,000 plt/ul) and individuals with von Willibrand's disease or other known platelet malfunction disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females >18 years of age undergoing esophagogastroduodenoscopy (EGD).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the number of patients achieving a VLE (volumetric laser endomicroscopy) image that includes stomach, gastro esophageal junction (GEJ) and esophagus. | 1 day
  Achieving a VLE image is defined as completing a full 6cm scan. This will be presented as a percentage of patients.

SECONDARY OUTCOMES:
The evaluation of procedural workflow and physician interface to the NvisionVLE Imaging Console. | 1 day
  Procedural workflow and physician interface to the console will be assessed by a questionnaire that will be completed by the investigational staff involved in the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Prashanthi Thota, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States